CLINICAL TRIAL: NCT00665639
Title: A Phase 3, Randomized, Double-Blind, Comparative Trial of Two Dosing Regimens of Micafungin (FK463) Versus Caspofungin for the Treatment of Esophageal Candidiasis
Brief Title: Trial of Two Dosing Regimens of Micafungin Versus Caspofungin for the Treatment of Esophageal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-7-008
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Candidiasis, Oral
Keywords: Micafungin; Esophageal Candidiasis; caspofungin
MeSH Terms: conditions — Candidiasis, Oral | interventions — Micafungin; Caspofungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): Daily dose
  Interventions: Drug: micafungin
- 2 (Active Comparator)
  Interventions: Drug: caspofungin
- 3 (Experimental): Every other day dose, alternating with placebo
  Interventions: Drug: micafungin

INTERVENTIONS:
Drug: micafungin — IV
  Other Names: Mycamine; FK463
  Arms: 1; 3
Drug: caspofungin — IV
  Arms: 2

SUMMARY:
To determine the efficacy and safety of daily doses of IV micafungin versus IV caspofungin for the treatment of esophageal candidiasis

ELIGIBILITY:
Inclusion Criteria:

* Esophageal candidiasis confirmed by endoscopy
* Negative pregnancy test for female patients of childbearing potential

Exclusion Criteria:

* Pregnant or nursing female patient
* Evidence of liver disease
* Another active opportunistic fungal infection and/or receiving acute systemic therapy for an opportunistic fungal infection
* Concomitant esophagitis caused by herpes simplex virus or cytomegalovirus
* Received an oral or topical antifungal agent within 48 hours or a systemic antifungal agent within 72 hours of first dose of study drug
* Known to be non-responsive to therapy in any prior systemic antifungal clinical trail
* Experienced > 2 episodes of esophageal candidiasis requiring systemic antifungal therapy
* History of anaphylaxis attributed to echinocandin class of antifungals

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2004-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Comparative incidence of success, defined as complete clearing of esophageal lesions | End of Therapy

SECONDARY OUTCOMES:
Overall therapeutic response | End of Therapy
Mycological response | End of Therapy
Clinical response | End of Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (31):
- Argentina (4):
  - 5 Sites, Buenos Aires
  - Córdoba
  - Neuquén
  - Santa Fe
- Brazil (8):
  - Barretos
  - 3 Sites, Belo Horizonte
  - Boqueirao-Santos
  - Campinas
  - 2 Sites, Curitiba
  - Nova Iguaçu
  - Parquelandia-Fortaleza
  - 7 Sites, São Paulo
- 4 Sites, Lima, Peru
- South Africa (18):
  - Gaborone, Botswana
  - Windoek, Nambia
  - Arcadia-Pretoria
  - Benoni
  - 2 Sites, Bloemfontein
  - Cape Town
  - Centurion
  - Dundee
  - Durban
  - Hatfield-Pretoria
  - Olifantsfontein
  - 2 Sites, Port Elizabeth
  - Potchefstroom
  - Pretoria
  - Pretoria West
  - Reiger Park
  - Richards Bay
  - Somerset West

REFERENCES:
- [Derived] Andes DR, Reynolds DK, Van Wart SA, Lepak AJ, Kovanda LL, Bhavnani SM. Clinical pharmacodynamic index identification for micafungin in esophageal candidiasis: dosing strategy optimization. Antimicrob Agents Chemother. 2013 Nov;57(11):5714-6. doi: 10.1128/AAC.01057-13. Epub 2013 Aug 19. PMID 23959319